CLINICAL TRIAL: NCT00495599
Title: Adipose Secretory Function in Patients Before & After Laparoscopic Surgery
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Vanderbilt University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 051215
Record Dates: First submitted 2007-07-02; First posted 2007-07-03 (Estimated); Last update posted 2016-11-21 (Estimated); Status verified 2016-11

CONDITIONS: Obesity
Keywords: Obese; Adipose Tissue; Visfatin; Gastric Bypass Surgery
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Cytokines assessed from fat tissue — Cytokines assessed from fat tissue

SUMMARY:
The central hypothesis of our study is that metabolic and hemodynamic improvements following gastric bypass surgery are mediated by downregulation of inflammation-related adipokines produced by the intra-abdominal adipose tissue such as Visfatin.

DETAILED DESCRIPTION:
Central obesity represents a major risk for the development of type 2 diabetes and cardiovascular complications. Obesity is often associated with insulin resistance and abnormal production of inflammatory cytokines. Adipose tissue and especially omentum (adipocytes and resident macrophages) release several cytokines. Visfatin corresponds to a protein identified previously as pre-B cell colony-enhancing factor (PBEF), a 52-kilodalton cytokine expressed in lymphocytes. [1] Visfatin exerted insulin-mimetic effects in cultured cells and lowered plasma glucose levels in mice. Mice heterozygous for a targeted mutation in the visfatin gene had modestly higher levels of plasma glucose relative to wild-type littermates. Surprisingly, visfatin binds to and activates the insulin receptor.

Adipose tissue protein and mRNA expression of Visfatin (PBEF) has not been investigated in a single study design with regard to the relationship to fat distribution, insulin resistance and other metabolic risk factors, especially in morbidly obese individual undergoing weight loss surgery. Therefore, we propose the following specific aims: Investigate the protein and mRNA expression of Visfatin (PBEF) in the peripheral (subcutaneous) and visceral (omentum) adipose tissues of morbidly obese subjects and their relationships to the changes in body composition, fat distribution, insulin sensitivity and time-dependent reversal of co-morbidities following gastric bypass surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a BMI < 35undergoing laparoscopic surgery;
* Patients undergoing bariatric surgery with a BMI >35kg/m2; and
* Those patients who have had gastric by-pass that require additional surgical procedures are eligible for this research protocol.

Exclusion Criteria:

* Unwilling to consent.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 107 (Actual)
Dates: Start 2006-03; Primary Completion 2009-11 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
The primary endpoint of the study is change in mRNA levels of Visfatin. | Levels of Visfatin will be assayed from fat tissue taken before and after gastric bypass surgery or other laparoscopic surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Alfonso Torquati, M.D., Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States